CLINICAL TRIAL: NCT03247452
Title: Impact of Low Fiber Diet on Colonic Cleansing Quality Prior to Colonoscopy: Randomized Study Comparing 1 Day Versus 3 Days of Low Fiber Diet
Brief Title: Impact of Low Fiber Diet on Colonic Cleansing Quality (DIETPREP)
Acronym: DIETPREP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario de Canarias (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Large bowel cleansing
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cleansing Quality of the Colon
Keywords: Low fiber diet; Colonoscopy; Bowel Cleansing
MeSH Terms: interventions — Polyethylene Glycols; Ascorbic Acid

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Only the endoscopists in charged of rating cleansing quality during colonoscopy will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- One-day low fiber diet (Active Comparator): Patients assigned to the active comparator will receive oral and written instructions about the same structured low fiber diet designed by an Endocrinologist but they will follow this diet only the day before colonoscopy.
  2 liters of polyethylene glycol plus ascorbic acid will be administered
  Interventions: Other: One-day Low fiber diet; Drug: Polyethylene Glycol plus ascorbic acid
- Three-day low fiber diet (Experimental): Patients assigned to the experimental group will receive oral and written instructions about a structured low fiber diet designed by an Endocrinologist. They must follow this diet three days before colonoscopy.
  2 liters of polyethylene glycol plus ascorbic acid will be administered
  Interventions: Other: Three-day low fiber diet; Drug: Polyethylene Glycol plus ascorbic acid

INTERVENTIONS:
Other: One-day Low fiber diet — One-day low fiber diet before colonoscopy
  Arms: One-day low fiber diet
Other: Three-day low fiber diet — Three days low fiber diet before colonoscopy
  Arms: Three-day low fiber diet
Drug: Polyethylene Glycol plus ascorbic acid — 2 liters of Polyethylene Glycol plus ascorbic acid will be administered to both groups

SUMMARY:
This is a single center randomized controlled trial to compare bowel cleansing for outpatient colonoscopy in two groups of participants: one group will receive instructions of one-day structured low fiber diet whilst the other group will receive three-day low fiber diet.

Both groups will receive the same bowel cleansing solution (polyethylene glycol plus ascorbic acid). Bowel cleansing will be assessed according the Boston Bowel Preparation Scale.

DETAILED DESCRIPTION:
It is well-known that low fiber diet before colonoscopy is at least equivalent to liquid diet. However, tolerance is better with low fiber diet. There is no current evidence whether the number of days on low fiber diet before colonoscopy have any influence on bowel cleansing quality.

This is the first controlled, randomized trial to compare bowel cleansing by using two different protocols: one day low fiber diet versus three day low fiber diet.

A researcher will offer to participate in the study to scheduled for outpatient colonoscopy, who meet all the inclusion criteria and none of the exclusion criteria. The researchers will explain the purpose of the study and will ask to sign the informed consent. They will give verbal and written information on the diet and the bowel cleansing solution to be taken. Thus, according to the allocation group, participants must comply with a low fiber diet the previous day of the examination or 3 days prior to the examination. In both cases, patients will take a liquid diet the night before.

Patients from both groups will receive low volume preparation with 1 L of polyethylene glycol plus ascorbic acid 12 hours prior to the appointment of the colonoscopy and 1 L of PEG with ascorbic acid 5 hours before the appointment for colonoscopy.

Patients must complete a baseline questionnaire at the inclusion visit and another questionnaire at the colonoscopy visit.

The hypothesis of the study is that in non-selected population, a 3-day low fiber diet before colonoscopy is superior to 1-day low fiber diet in achieving an acceptable bowel cleansing assessed by a validated scale (Boston Bowel Preparation Score).

For the present study, a 10% improvement in the quality of colonic cleaning was hypothesized in the group of patients receiving 3 day low fiber diet regimen. Taking into account a power of 80%, alpha error of 5% and losses of 15% will require 202 patients per group.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years

Exclusion Criteria:

* Patients with previous colon surgery
* Last colonoscopy with poor bowel preparation
* Ileus, intestinal obstruction, megacolon
* Poorly controlled hypertension (HTAS> 180 HTAD> 100)
* Terminal renal failure (pre-dialysis or dialysis)
* Congestive heart failure (NYHA III-IV)
* Acute liver failure
* Severe psychiatric illness
* Dementia with difficulty in the intake of the preparation
* Pregnancy or breastfeeding
* Phenylketonuria
* Deficiency of glucose-6-phosphate dehydrogenase
* Refusal to participate in the study
* Inability to follow the instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Boston Bowel Preparation Scale | 7 months
  This scale goes from 0 (no preparation) to 3 points (excellent preparation) in the three segments of the colon (Proximal, transverse and distal). Maximum punctuation is 9 points

SECONDARY OUTCOMES:
Proportion of polyps detected in each arm | 7 months
  Number of polyps detected in one arm/total of polyps detected
Degree of satisfaction with diet | 7 months
  It will be assessed using a visual scale (1 excellent to 10 unbearable)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Quintero, MD, PhD, Study Director — Hospital Universitario de Canarias
Locations (1):
- Department of Gastroenterology, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

REFERENCES:
- [Result] Hassan C, Bretthauer M, Kaminski MF, Polkowski M, Rembacken B, Saunders B, Benamouzig R, Holme O, Green S, Kuiper T, Marmo R, Omar M, Petruzziello L, Spada C, Zullo A, Dumonceau JM; European Society of Gastrointestinal Endoscopy. Bowel preparation for colonoscopy: European Society of Gastrointestinal Endoscopy (ESGE) guideline. Endoscopy. 2013;45(2):142-50. doi: 10.1055/s-0032-1326186. Epub 2013 Jan 18. PMID 23335011
- [Result] Song GM, Tian X, Ma L, Yi LJ, Shuai T, Zeng Z, Zeng XT. Regime for Bowel Preparation in Patients Scheduled to Colonoscopy: Low-Residue Diet or Clear Liquid Diet? Evidence From Systematic Review With Power Analysis. Medicine (Baltimore). 2016 Jan;95(1):e2432. doi: 10.1097/MD.0000000000002432. PMID 26735547
- [Result] Gimeno-Garcia AZ, Baute JL, Hernandez G, Morales D, Gonzalez-Perez CD, Nicolas-Perez D, Alarcon-Fernandez O, Jimenez A, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Carrillo M, Ramos L, Quintero E. Risk factors for inadequate bowel preparation: a validated predictive score. Endoscopy. 2017 Jun;49(6):536-543. doi: 10.1055/s-0043-101683. Epub 2017 Mar 10. PMID 28282690
- [Result] Wu KL, Rayner CK, Chuah SK, Chiu KW, Lu CC, Chiu YC. Impact of low-residue diet on bowel preparation for colonoscopy. Dis Colon Rectum. 2011 Jan;54(1):107-12. doi: 10.1007/DCR.0b013e3181fb1e52. PMID 21160321
- [Derived] Gimeno-Garcia AZ, de la Barreda Heuser R, Reygosa C, Hernandez A, Mascareno I, Nicolas-Perez D, Jimenez A, Lara AJ, Alarcon-Fernandez O, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Hernandez G, Hernandez D, Delgado R, Quintero E. Impact of a 1-day versus 3-day low-residue diet on bowel cleansing quality before colonoscopy: a randomized controlled trial. Endoscopy. 2019 Jul;51(7):628-636. doi: 10.1055/a-0864-1942. Epub 2019 Apr 3. PMID 30943553